CLINICAL TRIAL: NCT04834726
Title: Pragmatic Trial of COVID Vaccine Text Outreach Interventions
Brief Title: COVID-19 Vaccine Text Outreach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shivan J Mehta, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 848696
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: Vaccination Uptake; Text Messaging; Outreach
MeSH Terms: conditions — COVID-19 | interventions — Water Insecurity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- 1: Usual Care (Active Comparator): Patients will receive a phone call to schedule their appointment from an Access Center representative. Access Center representatives will make up to 3 attempts to schedule an appointment with the patient. Patients randomized to this arm will not receive any text messaging.
  Interventions: Behavioral: Phone Call
- 2A: Call Back + Standard Msg (Experimental): The message describes that the patient is eligible for the COVID vaccine. Will include a prompt to agree to scheduling. The access center will call these patients back to schedule, calling up to 3 times.
  Interventions: Behavioral: Opt-In (Call-Back); Behavioral: Standard Message
- 2B: Call Back + Clinician Endorsement (Experimental): The message will describe an endorsement from the provider to get the vaccination. Will include a prompt to agree to scheduling. The access center will call these patients back to schedule, calling up to 3 times.
  Interventions: Behavioral: Opt-In (Call-Back); Behavioral: Clinician Endorsement
- 2C: Call Back + Scarcity (Experimental): The message will highlight the limited availability and the elevated priority for the patient to receive the vaccine at Penn Medicine. Will include a prompt to agree to scheduling. The access center will call these patients back to schedule, calling up to 3 times.
  Interventions: Behavioral: Opt-In (Call-Back); Behavioral: Scarcity
- 2D: Call Back + Opt-Out Framing (Experimental): The message will highlight that a vaccine is reserved for the patient, implying that they need to opt-outWill include a prompt to agree to scheduling. The access center will call these patients back to schedule, calling up to 3 times.
  Interventions: Behavioral: Opt-In (Call-Back); Behavioral: Opt-Out Framing
- 3A: In-Bound Call + Standard Msg (Experimental): The message describes that the patient is eligible for the COVID vaccine. Will include a prompt to agree to scheduling, which will be followed by a prompt to call the Penn Medicine Vaccine Scheduling Hotline to schedule their vaccine appointment.
  Interventions: Behavioral: Opt-in (In-Bound); Behavioral: Standard Message
- 3B: In-Bound Call + Clinician Endorsement (Experimental): The message will describe an endorsement from the provider to get the vaccination. Will include a prompt to agree to scheduling, which will be followed by a prompt to call the Penn Medicine Vaccine Scheduling Hotline to schedule their vaccine appointment.
  Interventions: Behavioral: Opt-in (In-Bound); Behavioral: Clinician Endorsement
- 3C: In-Bound Call + Scarcity (Experimental): The message will highlight the limited availability and the elevated priority for the patient to receive the vaccine at Penn Medicine. Will include a prompt to agree to scheduling, which will be followed by a prompt to call the Penn Medicine Vaccine Scheduling Hotline to schedule their vaccine appointment.
  Interventions: Behavioral: Opt-in (In-Bound); Behavioral: Scarcity
- 3D: In-Bound Call + Opt-Out Framing (Experimental): The message will highlight that a vaccine is reserved for the patient, implying that they need to opt-out. Will include a prompt to agree to scheduling, which will be followed by a prompt to call the Penn Medicine Vaccine Scheduling Hotline to schedule their vaccine appointment.
  Interventions: Behavioral: Opt-in (In-Bound); Behavioral: Opt-Out Framing

INTERVENTIONS:
Behavioral: Opt-In (Call-Back) — Messaging will include a prompt to agree to scheduling. If patient agrees, the access center will call these patients back to schedule, calling up to 3 times.
  Arms: 2A: Call Back + Standard Msg; 2B: Call Back + Clinician Endorsement; 2C: Call Back + Scarcity; 2D: Call Back + Opt-Out Framing
Behavioral: Opt-in (In-Bound) — Messaging will include a prompt to agree to scheduling followed by a prompt to call the Penn Medicine Vaccine Scheduling Hotline to schedule their vaccine appointment.
  Arms: 3A: In-Bound Call + Standard Msg; 3B: In-Bound Call + Clinician Endorsement; 3C: In-Bound Call + Scarcity; 3D: In-Bound Call + Opt-Out Framing
Behavioral: Standard Message — The message describes that the patient is eligible for the COVID vaccine.
  Arms: 2A: Call Back + Standard Msg; 3A: In-Bound Call + Standard Msg
Behavioral: Clinician Endorsement — The message will describe an endorsement from the provider to get the vaccination.
  Arms: 2B: Call Back + Clinician Endorsement; 3B: In-Bound Call + Clinician Endorsement
Behavioral: Scarcity — The message will highlight the limited availability and the elevated priority for the patient to receive the vaccine at Penn Medicine.
  Arms: 2C: Call Back + Scarcity; 3C: In-Bound Call + Scarcity
Behavioral: Opt-Out Framing — This will highlight that a vaccine is reserved for the patient, implying that they need to opt-out.
  Arms: 2D: Call Back + Opt-Out Framing; 3D: In-Bound Call + Opt-Out Framing
Behavioral: Phone Call — The access center will call these patients to schedule their vaccine appointment. These patients will not receive text messaging.
  Arms: 1: Usual Care

SUMMARY:
This project aims to evaluate different approaches to increase COVID-19 vaccine uptake among at-risk patients at Penn Medicine in an equitable and systematic manner through a centralized outreach program. The investigators will evaluate different text-based scheduling and messaging approaches informed by behavioral science to increase uptake among eligible patients, including the use of clinician endorsement, opt-out framing, and scarcity.

DETAILED DESCRIPTION:
This project will evaluate a centralized approach to increasing COVID through direct outreach to eligible patients via text messaging. This pragmatic randomized controlled trial has the following aims:

Aim 1: To conduct systematic large scale text message outreach for vaccine delivery among a defined group of Penn Medicine in a way that advances equity.

Aim 2: To offer different scheduling workflows through text messaging that might increase uptake and reduce disparities.

Aim 3: To compare the equity and efficiency of different messages informed by behavioral science, including PCP endorsement, opt-out framing, and scarcity.

ELIGIBILITY:
Inclusion Criteria:

* patients of Penn Medicine aged 18+ who reside in Philadelphia and who have had at least 1 visit in the past 5 years with a Penn Medicine primary care provider (PCP)

Exclusion Criteria:

* Patients who have completed any dose of the vaccine at Penn Medicine, are currently scheduled to receive the vaccine, have externally documented vaccination records, or have previously received text-message based vaccine outreach.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19554 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Mallozzi C, Shaw PA, Reitz C, McDonald C, Vandertuyn M, Balachandran M, Kopinsky M, Sevinc C, Johnson A, Ward R, Park SH, Snider CK, Rosin R, Asch DA. Effect of Text Messaging and Behavioral Interventions on COVID-19 Vaccination Uptake: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2216649. doi: 10.1001/jamanetworkopen.2022.16649. PMID 35696165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Waiver of informed consent obtained. 19,554 patients randomized.
Period: Overall Study
Arm/Group | 1: Usual Care | 2A: Call Back + Standard Msg | 2B: Call Back + Clinician Endorsement | 2C: Call Back + Scarcity | 2D: Call Back + Opt-Out Framing | 3A: In-Bound Call + Standard Msg | 3B: In-Bound Call + Clinician Endorsement | 3C: In-Bound Call + Scarcity | 3D: In-Bound Call + Opt-Out Framing
Started | 472 | 2393 | 2389 | 2392 | 2385 | 2380 | 2382 | 2383 | 2378
Completed | 390 | 1971 | 1985 | 1977 | 1957 | 1918 | 1935 | 1934 | 1978
Not Completed | 82 | 422 | 404 | 415 | 428 | 462 | 447 | 449 | 400
Not completed — Excluded for receiving one or more vaccine doses prior to outreach | 82 | 422 | 404 | 415 | 428 | 462 | 447 | 449 | 400

BASELINE CHARACTERISTICS:
Population: All randomized patients who were not excluded from analyses for receiving one or more vaccine doses prior to outreach.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Usual Care | 2A: Call Back + Standard Msg | 2B: Call Back + Clinician Endorsement | 2C: Call Back + Scarcity | 2D: Call Back + Opt-Out Framing | 3A: In-Bound Call + Standard Msg | 3B: In-Bound Call + Clinician Endorsement | 3C: In-Bound Call + Scarcity | 3D: In-Bound Call + Opt-Out Framing | Total
Number analyzed (Participants) | 390 | 1971 | 1985 | 1977 | 1957 | 1918 | 1935 | 1934 | 1978 | 16045
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (11.6) | 36.7 (10.9) | 36.9 (10.6) | 36.9 (11.2) | 37.4 (11.6) | 36.7 (11.0) | 37.3 (11.2) | 36.7 (11.3) | 36.6 (10.9) | 36.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 235 | 1162 | 1193 | 1183 | 1115 | 1116 | 1105 | 1153 | 1156 | 9418
  Male | 155 | 809 | 792 | 794 | 842 | 802 | 830 | 781 | 822 | 6627
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 189 | 1040 | 1024 | 1023 | 1030 | 991 | 1017 | 1009 | 1022 | 8345
  Black | 127 | 568 | 597 | 598 | 575 | 563 | 550 | 553 | 575 | 4706
  Asian/Pacific Islander | 26 | 143 | 161 | 139 | 157 | 152 | 153 | 159 | 150 | 1240
  More Than One Race | 3 | 13 | 14 | 9 | 14 | 15 | 15 | 8 | 13 | 104
  Other Race | 45 | 207 | 189 | 208 | 181 | 197 | 200 | 205 | 218 | 1650
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 26 | 131 | 114 | 115 | 126 | 103 | 131 | 114 | 107 | 967
  Non-Hispanic/Latino | 352 | 1785 | 1824 | 1829 | 1800 | 1781 | 1761 | 1779 | 1815 | 14726
  Other Ethnicity | 12 | 55 | 47 | 33 | 31 | 34 | 43 | 41 | 56 | 352

OUTCOME MEASURES:

1. Primary Outcome: Dose 1 Completion
Description: Percentage of patients who complete the first dose of the COVID vaccine within 1 month of initial outreach
Time Frame: 1 month
Population: All randomized patients who were not excluded from analyses for receiving one or more vaccine doses prior to outreach.Comparisons were made between all patients assigned to a texting + outbound call arm (arms 2A+2B+2C+2D) and the outbound phone call only arm (arm 1), and between texting + inbound call arm (arms 3A+3B+3C+3D) and the outbound phone call only arm (arm 1). This was the original analysis as outlined in the protocol, which is why results are reported in this fashion.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Outbound Phone Only: Patients in this arm received a call from the patient vaccine access center to schedule a vaccine appointment.
- Arm 2: Text + Outbound Call: Patients in this arm received a text message asking if they would like to receive a call from the patient vaccine access center. Includes Arms 2A+2B+2C+2D
- Arm 3: Text + Inbound Call: Patients in this arm received a text asking if they would like to receive the phone number to call the patient access center to schedule their vaccine appointment. This arm includes 3A+3B+3C+3D.
Arm/Group | Arm 1: Outbound Phone Only | Arm 2: Text + Outbound Call | Arm 3: Text + Inbound Call
Number analyzed (Participants) | 390 | 7890 | 7765
Participants | 14 | 243 | 253

2. Secondary Outcome: Dose 1 Completion
Description: Percentage of patients who complete the first dose of the COVID vaccine within 2 months of initial outreach
Time Frame: 2 months
Population: All randomized patients who were not excluded from analyses for receiving one or more vaccine doses prior to outreach. Comparisons were made between all patients assigned to a texting + outbound call arm (arms 2A+2B+2C+2D) and the outbound phone call only arm (arm 1), and between texting + inbound call arm (arms 3A+3B+3C+3D) and the outbound phone call only arm (arm 1). This was the original analysis as outlined in the protocol, which is why results are reported in this fashion.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Outbound Phone Only | Arm 2: Text + Outbound Call | Arm 3: Text + Inbound Call
Number analyzed (Participants) | 390 | 7890 | 7765
Participants | 16 | 315 | 342

3. Secondary Outcome: Vaccine Completion
Description: Percentage of patients who complete the vaccination process within 2 months of initial outreach
Time Frame: 2 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Outbound Phone Only | Arm 2: Text + Outbound Call | Arm 3: Text + Inbound Call
Number analyzed (Participants) | 390 | 7890 | 7765
Participants | 13 | 222 | 231

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed.
Description: Adverse events were not monitored/assessed. The research solely tested methods of outreach for getting patients to complete the COVID vaccine, separately approved for use by the FDA with an EUA. No drug, medical device or medical procedure was under investigation.
Arm/Group | 1: Usual Care | 2A: Call Back + Standard Msg | 2B: Call Back + Clinician Endorsement | 2C: Call Back + Scarcity | 2D: Call Back + Opt-Out Framing | 3A: In-Bound Call + Standard Msg | 3B: In-Bound Call + Clinician Endorsement | 3C: In-Bound Call + Scarcity | 3D: In-Bound Call + Opt-Out Framing
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT04834726/Prot_SAP_000.pdf